CLINICAL TRIAL: NCT01766193
Title: Delivery Method and Risk for Urogenital Prolapse 15-20 Years Later
Acronym: uropro
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2012/666
Record Dates: First submitted 2013-01-07; First posted 2013-01-11 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Uterine Prolapse; Urinary Incontinence; Fecal Incontinence
Keywords: Delivery, obstetric; Obstetric Surgical Procedures; Vacuum Extraction, Obstetrical; Cesarean Section; Obstetrical Forceps; Epidemiology; Norway
MeSH Terms: conditions — Uterine Prolapse; Urinary Incontinence; Fecal Incontinence | interventions — Vacuum Extraction, Obstetrical; Cesarean Section

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- vaginal birth: women whose first child was born by spontaneous vaginal delivery
  Interventions: Procedure: vaginal delivery
- cesarean section: women whose first child was born by cesarean section
  Interventions: Procedure: cesarean section
- forceps: women whose first child was born by forceps extraction
  Interventions: Procedure: forceps extraction
- vacuum: women whose first child was born by vacuum extraction
  Interventions: Procedure: vacuum extraction

INTERVENTIONS:
Procedure: vaginal delivery
  Groups: vaginal birth
Procedure: forceps extraction — vaginal delivery by forceps extraction
  Groups: forceps
Procedure: vacuum extraction — vaginal delivery by vacuum extraction
  Groups: vacuum
Procedure: cesarean section
  Groups: cesarean section

SUMMARY:
The lifetime risk for a woman to undergo surgery for either vaginal prolapse or urinary incontinence is high. Previous studies have shown that pregnancy and childbirth are risk factors for developing prolapse. There is a lack of studies that follow women several years after delivery aiming to find whether symptoms of prolapse are linked to delivery method, ie vacuum, forceps, normal vaginal delivery and cesarean section. The investigators plan this study is to get more knowledge about pathology of prolapse and incontinence, to enable development of preventive strategies for these conditions.

Aim of the study is to determine whether the prevalence of symptoms and performed surgery for urogenital prolapse differs among women delivered by vacuum, forceps, normal vaginal delivery and cesarean section 15-20 years after their first delivery.

The investigators identify women that delivered their first child at St. Olavs Hospital, Trondheim, Norway between 1990-1997. Questionnaires will be sent to 2500 women (PFIQ-7, PFDI-20, PISQ-12), 600 of whom will get a clinical examination, where pelvic floor musculature is examined by palpation and 4D ultrasound, and a POP-Q quantification of prolapse performed.

ELIGIBILITY:
Inclusion Criteria:

* first delivery in time period 1990-1997
* vaginal birth, spontaneous, forceps or vacuum extraction, or cesarean section
* residency in Klæbu, Malvik, Melhus, Midtre Gauldal, Rissa, Selbu, Trondheim, Tydal, Åfjord at the time of first delivery

Exclusion Criteria:

* stillbirth
* breech birth
* congenital Abnormalities
* residency outside the 9 selected communities
* forceps delivery following previous vacuum extraction delivery or spontaneous vaginal birth
* vacuum extraction delivery following previous forceps delivery or spontaneous vaginal birth
* Vaginal birth following previous cesarean section

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women who delivered their first child at St. Olavs Hospital, Trondheim (Norway) between 1990-1997
Sampling Method: Non-Probability Sample
Enrollment: 1641 (Actual)
Dates: Start 2012-08; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
symptoms of urogenital prolapse | 15-20 years after first delivery
surgery for urogenital prolapse | 15-20 years after first delivery

SECONDARY OUTCOMES:
damage to pelvic floor musculature | 15-20 years after first delivery
urinary incontinence | 15-20 years after first delivery
anal incontinence | 15-20 years after first delivery

CONTACTS AND LOCATIONS:
Overall Officials: Kjell Å Salvesen, prof MD, Study Director — Norwegian University of Science and Technology; Siv Mørkved, PhD prof, Study Director — St. Olavs Hospital
Locations (1):
- St Olavs Hospital Trondheim University Hospital, Trondheim, Norway

REFERENCES:
- [Result] Volloyhaug I, Morkved S, Salvesen O, Salvesen K. Pelvic organ prolapse and incontinence 15-23 years after first delivery: a cross-sectional study. BJOG. 2015 Jun;122(7):964-71. doi: 10.1111/1471-0528.13322. Epub 2015 Feb 16. PMID 25683873
- [Result] Volloyhaug I, Morkved S, Salvesen O, Salvesen KA. Forceps delivery is associated with increased risk of pelvic organ prolapse and muscle trauma: a cross-sectional study 16-24 years after first delivery. Ultrasound Obstet Gynecol. 2015 Oct;46(4):487-95. doi: 10.1002/uog.14891. Epub 2015 Aug 25. PMID 25920322
- [Result] Volloyhaug I, Morkved S, Salvesen KA. Association between pelvic floor muscle trauma and pelvic organ prolapse 20 years after delivery. Int Urogynecol J. 2016 Jan;27(1):39-45. doi: 10.1007/s00192-015-2784-8. Epub 2015 Jul 22. PMID 26198007
- [Result] Volloyhaug I, Morkved S, Salvesen O, Salvesen KA. Assessment of pelvic floor muscle contraction with palpation, perineometry and transperineal ultrasound: a cross-sectional study. Ultrasound Obstet Gynecol. 2016 Jun;47(6):768-73. doi: 10.1002/uog.15731. Epub 2016 May 2. PMID 26300128